CLINICAL TRIAL: NCT04257006
Title: The Effects of oXiris on Systemic Inflammation, Endothelial Dysfunction and Volume Control in Cardiac Surgery Patients Undergoing Cardiopulmonary Bypass.
Brief Title: The Effects of Oxiris on Systemic Inflammation and Endothelial dysFunction
Acronym: EOSIEF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1BAX-2020
Record Dates: First submitted 2020-01-17; First posted 2020-02-05 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Acute Kidney Injury Due to Circulatory Failure (Disorder)
Keywords: acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients undergoing CRRT with oXiris membrane (Experimental): Elective cardiac surgery patients undergoing CPB we will range in 2 groups: I- with Prismaflex set oXiris (SCUF) after CPB, II- standard protocol.
  Indications for CRRT (SCUF) with oXiris after ICU admission:
  1. Signs of pulmonary edema after cardiac surgery, verified with X-ray control.
  Or high risk of pulmonary edema after cardiac surgery:
  1. Fluid overload ≥ 10%, measured with equation (%fluid overload= ((total fluid in- total fluid out)/admission body weight*100)
  2. CVP (central venous pressure) ˃ 12 mm H2O.
  3. PAWP (pulmonary arterial wedge pressure) ˃ 12 mm Hg, measured by Swan-Ganz catheter.
  In this arm the treatment of fluid overload will be provided via SCUF with oxiris membrane
  Interventions: Device: oXiris membrane
- standard protocol (No Intervention): Elective cardiac surgery patients undergoing CPB we will range in 2 groups: I- with Prismaflex set oXiris (SCUF) after CPB, II- standard protocol.
  Indications for CRRT (SCUF) with oXiris after ICU admission:
  1. Signs of pulmonary edema after cardiac surgery, verified with X-ray control.
  Or high risk of pulmonary edema after cardiac surgery:
  1. Fluid overload ≥ 10%, measured with equation (%fluid overload= ((total fluid in- total fluid out)/admission body weight*100)
  2. CVP (central venous pressure) ˃ 12 mm H2O.
  3. PAWP (pulmonary arterial wedge pressure) ˃ 12 mm Hg, measured by Swan-Ganz catheter.
  In this arm the management of fluid overload will be provided via diuretics or IHD (in condition diuretics treatment resistance)

INTERVENTIONS:
Device: oXiris membrane — Open heart surgery patients in early postoperative period with clinical signs of fluid overload undergoing CRRT
  Arms: patients undergoing CRRT with oXiris membrane

SUMMARY:
CS-AKI occurring in 20% to 70% of cases depending of the type of cardiac surgery. The systemic inflammatory response is often observed and associated with increased risk of AKI. Cardiopulmonary bypass (CPB) induces a complex inflammatory response that has a multifactorial pathogenesis. The inflammatory response is triggered by exposure of the blood to artificial surfaces during extracorporeal circulation, ischemia/reperfusion injuries, translocation of gram-negative bacteria from the intestinal tract, small amounts of LPS in IV solutions. SIRS during CPB with high levels of inflammatory mediators, active complement proteins and LPS provoke endothelial dysfunction- retraction of endothelial cells with increasing vascular permeability and thrombogenic activity, also inflammatory mediators activate leukocytes and they enhance vascular permeability by affecting endothelial cells and vascular basement membrane. The systemic inflammation and endothelial dysfunction are the basis for multiple organ dysfunction syndrome. Vascular integrity damage during cardiac surgery entail redistribution of fluids with interstitial fluid accumulation and require accurate volume control (pertinent removal of "CPB priming volume"), especially in patients with CKD (low GFR) with high risks of AKI.

DETAILED DESCRIPTION:
Specific details of Treatment/Intervention: (prescription and/or therapy, devices, equipment, solutions, product to be used in conducting study:

To apply Prismaflex system with oXiris membrane after cardiopulmonary bypass in SCUF modality for CPB priming volume elimination.

Duration of procedure: 6 hours Blood flow:150-200 ml/min Anticoagulation: no additional heparinization.

According to the features of oXiris membrane:

1. Cytokines, complement, endotoxin adsorptive capacity.
2. Capability of accurate fluid balance management after cardiac surgery and CPB.
3. Reduced demand of anticoagulation therapy for CRRT in patients with high risk of bleeding.

The goal of the research:

1. To evaluate effect of adsorption of oXiris membrane on levels of complement (C3a, C5a), pro- and anti-inflammatory cytokines (IL-1β, TNF-α,IL-6,Il-8, IL-10,TGF-β), LPS (EAA levels) after CPB.
2. To evaluate leukocytes activation after CPB and after inflammatory mediators adsorption with oXiris (CD11b/CD18)
3. To evaluate endothelial dysfunction after CPB and after CRRT with oXiris: endothelial/leukocytes interactions (ICAM-1, VCAM-1), biomarkers of endothelial permeability (angiopoetin-2, sFLT-1), biomarkers of endothelial coagulopathy (von Willebrand factor, thrombomodulin)
4. To evaluate effect of volume control with CRRT on CS-AKI and dependence on mechanical ventilation after cardiac surgery, regarding volume overload in patients undergoing CPB with "priming volume" infusion.
5. To evaluate stage and topography of cardiac surgery associated acute kidney injury (creatinine, cystatin C, NGAL, KIM-1, β2-microglobuline) in patients in two arms: oXiris and standard protocol.
6. To evaluate adsorptive and volume control feasible effects of oXiris membrane on volume management (CVP,PAWP), LPS adsorption, reduction of systemic inflammation , endothelium dysfunction and AKI after cardiac surgery with CPB in comparison with standard protocol.

ELIGIBILITY:
Inclusion Criteria:

* elective cardiac surgery patients undergoing CPB (>60 minutes) with valve replacement and CABG.

Exclusion Criteria:

* Immunosuppressive therapy, CKD 4 and 5 stages, RRT in last 90 days, pregnancy, autoimmune disease, allergy to heparin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Patient volume status assessment in perioperative period | in 24 hours
  To compare volume status in two arms based on CVP mmH2O and PAWP mmHg measurements

SECONDARY OUTCOMES:
survival after cardiac surgery | in 90 day
  to compare in arms with oxiris treatment and standard protocol amount of survived patients
'ICU and hospital length of stay after cardiac surgery. | in 28 days
  to compare in arms with oxiris treatment and standard protocol the amount of days spent in ICU wards and in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Yury Polushin, PhD, Principal Investigator — Pavlov First St. Petersburg State Medical University
Locations (1):
- Pavlov First St. Petersburg State Medical University, Saint Petersburg, Russsia, Russia

IPD SHARING:
Plan to Share IPD: Yes
de-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: data will be available within 1 year of study completion
Access Criteria: data access request will be reviewed by an external independent review panel.
URL: http://1spbgmu.ru